CLINICAL TRIAL: NCT04953351
Title: PROMUC Trial-Comparison of Magnetic Resonance Imaging-Ultrasound Fusion and Cognitive Registration in MR-targeted Prostate Biopsy: A Randomized Controlled Trial
Brief Title: MRI-Ultrasound Fusion or Cognitive Registration in MR-targeted Prostate Biopsy
Acronym: PROMUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MRITB-202003
Record Dates: First submitted 2021-07-01; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive registration targeted biopsy (Experimental)
  Interventions: Procedure: Cognitive registration targeted biopsy and TRUS-system biopsy
- MRI-ultrasound fusion targeted biopsy (Active Comparator)
  Interventions: Procedure: MRI-ultrasound fusion targeted biopsy and TRUS-system biopsy

INTERVENTIONS:
Procedure: Cognitive registration targeted biopsy and TRUS-system biopsy — Cognitive registration is a visual guidance technique in which the surgeon samples a visually estimated location on ultrasound that corresponds to the MRI suspicious regions location. TRUS-system biopsy includes 12 biopsy cores.
  Arms: cognitive registration targeted biopsy
Procedure: MRI-ultrasound fusion targeted biopsy and TRUS-system biopsy — MRI-ultrasound fusion targeted biopsy is conducted with an mpMRI-TRUS biopsy system that provides realtime fusion of TRUS images and MRI images to guide the biopsy needles. TRUS-system biopsy includes 12 biopsy cores.
  Arms: MRI-ultrasound fusion targeted biopsy

SUMMARY:
This randomized controlled trial aims to assess the detection rate of clinically significant and clinically insignificant cancer of MRI-ultrasound fusion targeted biopsy compared to cognitive registration targeted biopsy in men with clinical suspicion of prostate cancer who had no prior prostate biopsy.

DETAILED DESCRIPTION:
Prostate biopsy with multiple samples using a standardized template (standard biopsy, SB) under transrectal ultrasound (TRUS) guidance is the current standard diagnostic approach in suspicion of prostate cancer (PCa). However, many biopsies are unnecessary or cannot detect clinically significant PCa (csPCa).

With the introduction of multiparametric magnetic resonance imaging (mpMRI) of the prostate and the improvement for PCa detection and localization, an alternative procedure, known as MRI-targeted biopsy (MRI-TB), has been shown comparable or even higher detection rates of csPCa compared to TRUS-system biopsy (SB). MRI-ultrasound fusion TB (FUS-TB) and cognitive registration TB (COG-TB) are two techniques of MRI-TB commonly used. However, the optimal methodology for targeting MRI-suspicious regions remains unknown. The accuracy of COG-TB compared with FUS-TB remains unclear.

This randomized controlled trial aims to assess the detection rate of clinically significant and clinically insignificant cancer of COG-TB compared to FUS-TB (transperineal) in men referred with clinical suspicion of prostate cancer who have had no prior prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Men more than 18 years old with clinical suspicion of prostate cancer;
2. Serum PSA ≤ 20 ng/ml within the previous 3 months;
3. Suspected stage ≤ T2 on rectal examination (organ-confined prostate cancer) within the previous 3 months;
4. No evidence of PSA increase by noncancerous factors, such as catheterization, bladder stones, or urinary tract infection including bacterial prostatitis;
5. mpMRI PI-RADS V2.1 score ≥3；
6. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy or prostate surgery;
2. Prior treatment for prostate cancer;
3. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated glomerular filtration rate ≤ 50mls/min);
4. Contraindication to prostate biopsy;
5. Men in whom artifact would reduce the quality of the MRI.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Detection rates of clinically significant PCa in FUS-TB and COG-TB | When histology results available, at an expected average of 30 days post-biopsy

SECONDARY OUTCOMES:
Detection rates of clinically insignificant PCa in FUS-TB and COG-TB | When histology results available, at an expected average of 30 days post-biopsy
Detection rates of clinically insignificant PCa in men with MRI score 3, 4 or 5 | When histology results available, at an expected average of 30 days post-biopsy
Cancer core length of the most involved biopsy core (maximum cancer core length) | When histology results available, at an expected average of 30 days post-biopsy
Biopsy-related adverse events | 30 days post biopsy
Proportion of men undergoing radical prostatectomy who have Gleason grade upgrading | 60 days post biopsy
Detection rates of clinically significant PCa in SB | When histology results available, at an expected average of 30 days post-biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Guo, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China